CLINICAL TRIAL: NCT02451579
Title: A Randomized, Double-blind, Placebo-controlled, Prospective Clinical Trial Evaluating the Role of Systemic Antihistamine Therapy in the Reduction of Adverse Effects Associated With Topical 5-aminolevulinic Acid Photodynamic Therapy
Brief Title: A Clinical Trial Evaluating the Role of Systemic Antihistamine Therapy in the Reduction of Adverse Effects Associated With Topical 5-aminolevulinic Acid Photodynamic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDT-2015-01
Record Dates: First submitted 2015-05-12; First posted 2015-05-22 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratoses; Photodynamic Therapy; PDT; Blue Light
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetirizine Hydrochloride (Active Comparator): Prophylactic use of cetirizine hydrochloride prior to and after Topical 5-aminolevulinic Acid Photodynamic Therapy
  Interventions: Drug: Antihistamine Cetirizine Hydrochloride
- Placebo (Placebo Comparator): Prophylactic use of placebo prior to and after Topical 5-aminolevulinic Acid Photodynamic Therapy
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Antihistamine Cetirizine Hydrochloride — Prophylactic use of antihistamine prior to and following topical 5-aminolevulonic acid photodynamic therapy
  Arms: Cetirizine Hydrochloride
Other: Placebo — Use of placebo prior to and following topical 5-aminolevulonic acid photodynamic therapy
  Arms: Placebo

SUMMARY:
A double-blind, placebo controlled study conducted at a single study site. Evaluating the role of systemic antihistamine therapy in the reduction of adverse effects associated with topical 5-aminolevulinic acid photodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Subjects with 5-20 actinic keratosis of the face
* Patients undergoing photodynamic therapy (PDT) to the face for AK with 5-aminolevulinic acid (ALA) activated by blue light.
* Must be willing to give and sign a HIPPA form, photo consent and informed consent form.
* Must be willing to comply with study dosing and complete the entire course of the study.
* Female patients will be either of non-childbearing potential defined as:

  1. Having no uterus
  2. No menses for at least 12 months.

Or;

(WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as:

1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
2. Intrauterine coil
3. Bilateral tubal ligation
4. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
5. Abstinence (If practicing abstinence must agree to use barrier method described above (d) if becomes sexually active).
6. Vasectomized partner g. Negative urine pregnancy test results Baseline prior to study entry (if applicable)

Exclusion Criteria:

* Presence of incompletely healed wound in treatment area
* Presence of known or suspected BCC or SCC in treatment area
* Previous PDT or treatment of the face with any topical cytotoxic or immunomodulatory agent for AKs within the past 6 months
* Co-existing potentially confounding skin condition within treatment area (e.g. eczema, psoriasis, XP, rosacea) at investigator's discretion
* Presence of tattoo and/or scar in the treatment area that in the investigators opinion would interfere with study assessments
* Subjects with known photosensitivity or taking photosensitizing medications listed below:

  1. Oral diabetes medicines
  2. Griseofulvin
  3. Thiazide diuretics
  4. Sulfonylureas
  5. Phenothiazines
  6. Tetracycline's
  7. St. John's Wort
* Use of oral/topical retinoids within 1 month of Baseline
* Subjects with a history of sensitivity to porphyrins
* Subjects with recently excessive exposure of the treatment area to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of tanning during the time of the study
* Female subjects who are pregnant, nursing an infant or planning a pregnancy during the study [throughout the course of the study
* Presence or evidence of any conditions that in the opinion of the investigator might impede the subject's ability to give consent or comply with protocol requirements.
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study
* History of non-compliance with clinical research protocols
* Ablative laser resurfacing to on their face within 12 months
* Non-ablative laser or light procedures to their face within the past 3 months
* Microdermabrasion (light or medium skin peel) treatment on their face within the past 30 days

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Localized Skin Response | Up to day 180
  Localized Skin Response consisting of erythema, edema, crusting, exudation, Vesiculation/Pustulation and erosion/ ulceration Investigator evaluated on a standardized scale

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States

REFERENCES:
- [Derived] Vanaman Wilson MJ, Jones IT, Wu DC, Goldman MP. A randomized, double-blind, placebo-controlled clinical trial evaluating the role of systemic antihistamine therapy for the reduction of adverse effects associated with topical 5-aminolevulinic acid photodynamic therapy. Lasers Surg Med. 2017 Oct;49(8):738-742. doi: 10.1002/lsm.22682. Epub 2017 May 10. PMID 28489298